CLINICAL TRIAL: NCT03246958
Title: A Phase 2 Study of Nivolumab Plus Ipilimumab in RAI Refractory, Aggressive Thyroid Cancer With Exploratory Cohorts in Medullary and Anaplastic Thyroid Cancer
Brief Title: Nivolumab Plus Ipilimumab in Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Kartik Sehgal, MD, Kartik Sehgal, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-255
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- DTC - Nivolumab alone for two weeks (Experimental): Differentiated Thyroid Cancer (DTC) participants received Ipilimumab 1mg/kg q6 weeks via IV infusion, starting two weeks after Nivolumab 3mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- DTC - Ipilimumab alone for two weeks (Experimental): Differentiated Thyroid Cancer (DTC) participants received Nivolumab 3mg/kg q6 weeks via IV infusion, starting two weeks after Ipilimumab 1mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Differentiated Thyroid Cancer (Primary cohort) (Experimental): Differentiated Thyroid Cancer (DTC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second.
  Per protocol order in sequential design was not expected to impact efficacy rather was for exploratory correlative analyses. Participants were treated indefinitely until disease progression or withdrawal for other reasons.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Medullary Thyroid Cancer (Exploratory Cohort) (Experimental): Medullary Thyroid Cancer (MTC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second, or started Ipi or Nivo together.
  Per protocol order in sequential design was not expected to impact efficacy rather was for exploratory correlative analyses. Participants were treated indefinitely until disease progression or withdrawal for other reasons.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Anaplastic Thyroid Cancer (Exploratory Cohort) (Experimental): Anaplastic Thyroid Cancer (ATC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second prior to study amendment or in combination from the start after study amendment due to aggressive nature of the disease in this cohort.
  Per protocol order in sequential design was not expected to impact efficacy rather was for exploratory correlative analyses. Participants were treated indefinitely until disease progression or withdrawal for other reasons.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- MTC - Nivolumab alone for two week (Experimental): Medullary Thyroid Cancer (MTC)participants received Ipilimumab 1mg/kg q6 weeks via IV infusion, starting two weeks after Nivolumab 3mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- MTC - Ipilimumab alone for two weeks (Experimental): Medullary Thyroid Cancer (MTC) participants received Nivolumab 3mg/kg q6 weeks via IV infusion, starting two weeks after Ipilimumab 1mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ATC - Nivolumab alone for two week (Experimental): Anaplastic Thyroid Cancer (ATC) received Ipilimumab 1mg/kg q6 weeks via IV infusion, starting two weeks after Nivolumab 3mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ATC - Ipilimumab alone for two week (Experimental): Anaplastic Thyroid Cancer (ATC) received Nivolumab 3mg/kg q6 weeks via IV infusion, starting two weeks after Ipilimumab 1mg/kg q6 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- ATC - Ipilimumab + Nivolumab (Experimental): Anaplastic Thyroid Cancer (ATC) received Nivolumab 3mg/kg q6 weeks and Ipilimumab 1mg/kg q6 weeks via IV infusion.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Ipilimumab are types of immunotherapy Immunotherapy works by encouraging the body's own immune system to attack cancer cells.
  Other Names: Opdivo
Drug: Ipilimumab — Nivolumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells.
  Other Names: Yervoy

SUMMARY:
This research study is studying nivolumab, an investigational drug, in combination with ipilimumab, also an investigational drug, as a possible treatment for thyroid cancer.

The drugs involved in this study are:

* Nivolumab (Opdivo™)
* Ipilimumab (Yervoy™)

DETAILED DESCRIPTION:
This research study is a Phase 2 clinical trial. Phase 2 clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The purpose of this study is to evaluate effectiveness (how well the drug/s work) of nivolumab combined with ipilimumab.

Nivolumab and ipilimumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack cancer cells. Nivolumab has been approved by the US Food and Drug Administration (FDA) for the treatment of metastatic melanoma (a type of skin cancer), and specific types of previously treated advanced lung and kidney cancers. Ipilimumab is approved by the FDA for the treatment of metastatic melanoma.

The combination of nivolumab and ipilimumab is now FDA approved as treatment for patients with metastatic melanoma. However, the use of nivolumab as well as ipilimumab alone or in combination for the treatment of patients with thyroid cancer is not approved

ELIGIBILITY:
Inclusion

* Metastatic, RAI refractory, differentiated thyroid cancer (including papillary and follicular thyroid cancer and their sub-types such as Hurthle cell thyroid cancer as well as poorly differentiated thyroid cancer), with progression within 13 months prior to study registration. RAI refractoriness is defined as absence of uptake of RAI on either a low-dose diagnostic test or a post-treatment RAI scan in measurable lesions or radiographic progression of disease within 12 months of the last course of RAI treatment despite the recorded uptake of RAI with that previous therapy or having a cumulative lifetime administered dose of greater than 600mCi.
* Exploratory cohort: incurable medullary thyroid cancer with prior tyrosine kinase inhibitor (TKI) failure and progression within 13 months prior to enrollment (10 patients) and anaplastic thyroid cancer (7 patients)
* Any number of lines of prior treatment are allowed
* Any line of prior treatment for patients under 65y, over 65y must have at least one prior line of TKI treatment
* Age 18 years or older
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:
* Screening laboratory values must meet the following criteria and should be obtained within 21 days prior to randomization/registration

  * WBC ≥ 2000/μL
  * Neutrophils ≥ 1500/μL
  * Platelets ≥ 100 x103/μL
  * Hemoglobin > 9.0 g/dL
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
  * AST/ALT ≤ 3 x ULN
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Ability to understand and the willingness to sign a written informed consent document.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 iu/l or equivalent units of hcg) within 24 hours of the first dose of the study drug
* Women of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception

Exclusion

* Patients should be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with activebrain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sehgal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sehgal K, Pappa T, Shin KY, Schiantarelli J, Liu M, Ricker C, Besson NR, Jones SM, Welsh EL, Pfaff KL, Barletta JA, Park J, Reardon B, Doherty GM, Alexander EK, Rodig SJ, Barbie DA, O'Neill A, Van Allen E, Haddad RI, Lorch JH. Dual Immune Checkpoint Inhibition in Patients With Aggressive Thyroid Carcinoma: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2024 Dec 1;10(12):1663-1671. doi: 10.1001/jamaoncol.2024.4019. PMID 39446365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from October 2017 to July 2019.
Pre-assignment Details: Per protocol order in sequential design was not expected to impact efficacy rather was for exploratory correlative analyses.
Groups:
- MTC - Nivolumab Alone for Two Week: Medullary Thyroid Cancer (MTC) participants received Ipilimumab 1mg/kg q6 weeks via IV infusion, starting two weeks after Nivolumab 3mg/kg q6 weeks.
Period: Overall Study
Arm/Group | DTC - Nivolumab Alone for Two Weeks | DTC - Ipilimumab Alone for Two Weeks | MTC - Nivolumab Alone for Two Week | MTC - Ipilimumab Alone for Two Weeks | ATC - Nivolumab Alone for Two Week | ATC - Ipilimumab Alone for Two Week | ATC - Ipilimumab + Nivolumab
Started | 17 | 18 | 3 | 4 | 2 | 4 | 4
Analyzable | 16 | 16 | 3 | 4 | 2 | 4 | 4
Completed | 1 | 3 | 0 | 0 | 0 | 1 | 1
Not Completed | 16 | 15 | 3 | 4 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Progression | 13 | 9 | 3 | 2 | 1 | 2 | 1
Not completed — Adverse Event | 2 | 2 | 0 | 1 | 1 | 0 | 2
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Never start treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Over enrollment | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is the subset of patients that were analyzable.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTC - Nivolumab Alone for Two Weeks | DTC - Ipilimumab Alone for Two Weeks | MTC - Nivolumab Alone for Two Week | MTC - Ipilimumab Alone for Two Weeks | ATC - Nivolumab Alone for Two Week | ATC - Ipilimumab Alone for Two Week | ATC - Ipilimumab + Nivolumab | Total
Number analyzed (Participants) | 16 | 16 | 3 | 4 | 2 | 4 | 4 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.9 (11.8) | 63.4 (10.3) | 54.7 (2.9) | 51.8 (16.3) | 51.4 (2.1) | 69.3 (16.9) | 58.4 (8.3) | 62.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 2 | 2 | 0 | 4 | 2 | 25
  Male | 8 | 9 | 1 | 2 | 2 | 0 | 2 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 16 | 15 | 2 | 4 | 2 | 3 | 4 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 15 | 0 | 2 | 0 | 0 | 0 | 3 | 20
  Asian | 1 | 15 | 0 | 4 | 2 | 3 | 0 | 25
  Other | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) PS: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out of work of a light or sedentary nature (PS2) Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about >50% of waking hours
  Participants
    0 | 6 | 6 | 0 | 1 | 0 | 3 | 1 | 17
    1 | 9 | 8 | 3 | 3 | 2 | 3 | 3 | 31
    2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: Best overall response rate is defined as the percentage of participants who achieved Complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Median (range) treatment duration (days) of 163.0 (21.0-734.0) for DTC cohort, for MTC cohort was 58.0 (30.0-252.0), and for ATC cohort 135.5 (10.0-735.0).
Population: It was pre-specified in the Study Protocol to report data by disease cohort irrespective of assigned treatment sequence.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Differentiated Thyroid Cancer (Primary Cohort): Differentiated Thyroid Cancer (DTC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second.
  Participants were treated indefinitely until disease progression or withdrawal for other reasons.
- Medullary Thyroid Cancer (Exploratory Cohort): Medullary Thyroid Cancer (MTC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second.
  Participants were treated indefinitely until disease progression or withdrawal for other reasons.
- Anaplastic Thyroid Cancer (Exploratory Cohort): Anaplastic Thyroid Cancer (ATC) participants received Ipilimumab (Ipi) 1mg/kg q6 weeks and Nivolumab (Nivo) 3mg/kg q6 weeks sequentially either Ipi or Nivo first with 2 weeks apart prior to start of either Ipi or Nivo second prior to study amendment or in combination from the start after study amendment due to aggressive nature of the disease in this cohort.
  Participants were treated indefinitely until disease progression or withdrawal for other reasons.
Arm/Group | Differentiated Thyroid Cancer (Primary Cohort) | Medullary Thyroid Cancer (Exploratory Cohort) | Anaplastic Thyroid Cancer (Exploratory Cohort)
Number analyzed (Participants) | 32 | 7 | 10
percentage of participants | 9.4 [2.8 to 28.5] | 0 [0 to 41] | 30 [6.7 to 65.2]

2. Secondary Outcome: Median Progression Free Survival
Description: Progression-Free Survival (PFS) based on Kaplan-Meier methodology is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Median (range) follow-up (months) for DTC cohort was 24.0 (1.84 - 24.7), for MTC cohort was 24.0 (23.0-24.2), and for ATC cohort was 22.2 (0.46 - 26.1).
Population: It was pre-specified in the Study Protocol to report data by disease cohort irrespective of assigned treatment sequence.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Differentiated Thyroid Cancer (Primary Cohort) | Medullary Thyroid Cancer (Exploratory Cohort) | Anaplastic Thyroid Cancer (Exploratory Cohort)
Number analyzed (Participants) | 32 | 7 | 10
Months | 7.11 [2.07 to 17.02] | 2.14 [0.92 to 3.98] | 4.29 [0.46 to NA] — NA due to limited number of events.

3. Secondary Outcome: Overall Survival at 2 Years (OS2)
Description: Overall Survival is the percent probability estimate at 2 years based on Kaplan-Meier methodology. OS is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Time Frame: as for outcome 2
Population: It was pre-specified in the Study Protocol to report data by disease cohort irrespective of assigned treatment sequence.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Differentiated Thyroid Cancer (Primary Cohort) | Medullary Thyroid Cancer (Exploratory Cohort) | Anaplastic Thyroid Cancer (Exploratory Cohort)
Number analyzed (Participants) | 32 | 7 | 10
Percent Probability | 77.2 [58.1 to 88.5] | 85.7 [33.4 to 97.9] | 55.6 [20.4 to 80.5]

4. Secondary Outcome: Treatment-Related Adverse Events Rate
Description: Treatment-related adverse events rate was defined as the proportion of participants who experienced an adverse event with treatment attribution of possible, probable or definite, including all grades based on the Common Toxicity Criteria for Adverse Events Version 4.0 (CTCAEv4) as reported on case report forms.
Time Frame: AEs were assessed every two weeks on treatment and within 30 days after the last dose. Median (range) treatment duration (days) of 163.0 (21.0-734.0) for DTC cohort, for MTC cohort was 58.0 (30.0-252.0), and for ATC cohort 135.5 (10.0-735.0).
Population: It was pre-specified in the Study Protocol to report data by disease cohort irrespective of assigned treatment sequence.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Differentiated Thyroid Cancer (Primary Cohort) | Medullary Thyroid Cancer (Exploratory Cohort) | Anaplastic Thyroid Cancer (Exploratory Cohort)
Number analyzed (Participants) | 32 | 7 | 10
proportion of participants | 0.81 [0.64 to 0.93] | 1 [0.59 to 1] | 0.80 [0.44 to 0.97]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every two weeks while participants were on treatment and within 30 days after the last dose. Participants at DTC cohort received a median treatment duration of 163.0 days (range 21.0-734.0), for MTC cohort 58.0 days (range 30.0 - 252.0), and for ATC cohort 135.5 days (range 10.0 - 735.0). For death, median follow-up for DTC cohort was 24.0 months (range 1.84 - 24.7), for MTC cohort 24.0 months (range 23.0-24.2), and for ATC cohort 22.2 months (range 0.46 - 26.1).
Description: SAE defined as any expected or unexpected adverse event, related or unrelated to the therapy being studied, occurring at any agent dose, any phase of product, or procedure testing, that results in any of the following outcomes:death, a life-threatening adverse event requires inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity new cancer, congenital anomaly or birth defect. All others were OAEs.
Arm/Group | DTC - Nivolumab Alone for Two Weeks | DTC - Ipilimumab Alone for Two Weeks | MTC - Nivolumab Alone for Two Week | MTC - Ipilimumab Alone for Two Weeks | ATC - Nivolumab Alone for Two Week | ATC - Ipilimumab Alone for Two Week | ATC - Ipilimumab + Nivolumab
All-Cause Mortality (participants affected / at risk) | 5/16 | 5/16 | 1/3 | 0/4 | 1/2 | 2/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 5/16 | 3/16 | 1/3 | 0/4 | 2/2 | 2/4 | 0/4
Other Adverse Events (participants affected / at risk) | 16/16 | 16/16 | 3/3 | 4/4 | 2/2 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTC - Nivolumab Alone for Two Weeks (N=16) | DTC - Ipilimumab Alone for Two Weeks (N=16) | MTC - Nivolumab Alone for Two Week (N=3) | MTC - Ipilimumab Alone for Two Weeks (N=4) | ATC - Nivolumab Alone for Two Week (N=2) | ATC - Ipilimumab Alone for Two Week (N=4) | ATC - Ipilimumab + Nivolumab (N=4)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTC - Nivolumab Alone for Two Weeks (N=16) | DTC - Ipilimumab Alone for Two Weeks (N=16) | MTC - Nivolumab Alone for Two Week (N=3) | MTC - Ipilimumab Alone for Two Weeks (N=4) | ATC - Nivolumab Alone for Two Week (N=2) | ATC - Ipilimumab Alone for Two Week (N=4) | ATC - Ipilimumab + Nivolumab (N=4)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 2 | 1 | 1 | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 7 | 1 | 2 | 0 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 4 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 7 | 0 | 2 | 1 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 5 | 5 | 1 | 0 | 0 | 1 | 1
Edema trunk (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 8 | 1 | 2 | 2 | 2 | 0
Fever (General disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 1
Flu like symptoms (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 5 | 5 | 1 | 2 | 1 | 2 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 3 | 3 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 5 | 5 | 2 | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 2 | 2 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 5 | 1 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 3 | 0 | 1 | 0 | 0 | 0
Cholesterol high (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 5 | 5 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 5 | 5 | 1 | 2 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Serum amylase increased (Investigations) | 4 | 4 | 0 | 1 | 0 | 1 | 1
Weight loss (Investigations) | 1 | 1 | 2 | 0 | 1 | 0 | 0
Investigations - Other, specify (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 5 | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 5 | 0 | 3 | 1 | 1 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 1 | 0 | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 1 | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 6 | 0 | 1 | 0 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 1 | 0 | 1 | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 2
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 4 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Limited number of patients accrued into ATC and MTC cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03246958/Prot_SAP_000.pdf